CLINICAL TRIAL: NCT01996618
Title: Reduction of Symptomatic Ventricular Premature Beats With Ranolazine
Brief Title: Study to Reduce Symptoms of Premature Beats With Ranolazine
Acronym: RSVP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20043-7
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2013-11

CONDITIONS: Premature Ventricular Beats
Keywords: Premature Ventricular Beats; Premature Heart Beats; Ranolazine
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Experimental): Subjects will be consented by the study investigator and then randomly assigned in an allocation-concealed fashion to double blinded treatment with either titrated doses of ranolazine or matched placebo. After the initial 6 days of treatment with ranolazine, 500 mg twice daily or matched placebo, subjects will undergo repeat 24 hour electrocardiographic monitoring. If tolerated, the subjects will then have their study medication increased (Ranolazine 1,000 mg twice daily or matching placebo) with the plan to then undergo a repeat 24 hour ambulatory electrocardiographic monitoring in 6 days. When the subject returns the monitor, subjects will enter the washout period (cessation of the study medication) for 6 days and have electrocardiographic monitoring prior to return to the subject's referring provider for care.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Subjects will be consented by the study investigator and then randomly assigned in an allocation-concealed fashion to double-blinded treatment with either titrated doses of ranolazine or matched placebo. After the initial 6 days of treatment with ranolazine, 500 mg twice daily or matched placebo, subjects will undergo repeat 24 hour electrocardiographic monitoring. If tolerated, the subjects will then have their study medication increased (Ranolazine 1,000 mg twice daily or matching placebo) with the plan to then undergo a repeat 24-hour ambulatory electrocardiographic monitoring in 6 days. When the subject returns the monitor, subjects will enter the washout period (cessation of the study medication) for 6 days and have electrocardiographic monitoring prior to return to the subject's referring provider for care.

INTERVENTIONS:
Drug: Ranolazine — After the initial 6 days of treatment with ranolazine, 500 mg twice daily or matched placebo, subjects will undergo repeat 24 hour electrocardiographic monitoring. If tolerated, the subjects will then have their study medication increased (Ranolazine 1,000 mg twice daily) with the plan to then undergo a repeat 24 hour ambulatory electrocardiographic monitoring in 6 days.
  Other Names: Ranexa
  Arms: Ranolazine

SUMMARY:
Investigate whether ranolazine, a novel anti-anginal agent with antiarrhythmic properties, has a role in the management of symptomatic ventricular premature beats.

DETAILED DESCRIPTION:
The main objective is to compare the effect of ranolazine versus placebo on premature ventricular beats (using 24-hour ambulatory electrocardiographic monitoring) for subjects with symptomatic palpitations. Subject population will consist of seventy-two adult subjects of both sexes who have greater than 1,000 premature ventricular beats during initial monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female 18 years and older
* Symptoms of palpitations
* Greater than or equal to 1,000 Ventricular Premature Beats during 24-hour electrocardiographic monitoring
* Completion of a consent form prior to pre-randomization Holter monitor

Exclusion Criteria:

* Moderate to severe symptomatic heart failure, New York Heart Association Class III/IV
* Moderate to severe symptomatic angina, Canadian Cardiovascular Classification III/IV
* Moderate to severe structural heart disease in the absence of an implantable cardiac defibrillator in a subject who would otherwise be eligible for a defibrillator (e.g. history of myocardial infarction and a left ventricular ejection fraction less than 30%)
* Clinically significant hepatic disease (cirrhosis or chronic hepatitis) or abnormal liver associated enzymes greater than three times the upper limits of normal
* A baseline corrected QT interval greater than or equal to 500msec or history of congenital channelopathy (long QT syndrome, Brugada syndrome) or torsades de pointes.
* Treatment with agents known to prolong the QTc interval
* Treatment with agents that are potent or moderately potent inhibitors of CYP3A, to include, but is not limited to the following: ketoconazole, HIV protease inhibitors (i.e. ritonavir), macrolide antibiotics (i.e. clarithromycin), diltiazem and verapamil
* Females who are pregnant, planning to get pregnant, or breast feeding ( females under the age of 55 years who have not previously undergone surgical sterilization procedures will have serum qualitative pregnancy testing)
* Thyroid stimulating hormone less than 0.27 IU/mL
* Serum magnesium less than 1.5mg/dL
* Serum potassium less than 3.5 mEq/dL or greater than 5.0 mEq/dL
* Estimated GFR less than 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in Premature Ventricular Beats | 24-hour Holter Monitor after 14 days of therapy
  The primary endpoint will be a 50% reduction in premature ventricular beats during 24-hour Holter monitoring after randomization to active treatment or placebo for 14 days of therapy.

SECONDARY OUTCOMES:
Changes in transthoracic echocardiographic parameters | 14 days of therapy
  Measure changes in transthoracic echocardiographic parameters including diastolic parameters, mitral inflow velocities and deceleration time and mitral annular velocities using tissue doppler imaging.
Frequency of palpitations | 14 days of therapy
  Patient perceived change in frequency of palpitations from baseline to follow-up visit.
Reduction of Premature Atrial Beats | 24-hour Holter Monitor after 14 days of therapy
  Reduction of premature atrial beats during 24-hour holter monitoring after randomization to active treatment or placebo following 14 days of therapy.
Measure Temperature Rebound Rate (TRR) | 14 days of therapy
  Measure serial change in endothelial function as measured using the Vendys® DTM device as measured by fingertip Temperature Rebound (TR) in degrees Celsius. Temperature rebound is measured as the absolute difference between low fingertip temperature during cuff occlusion and maximal temperature rebound following cuff release. In addition, rate of change (slope) in temperature rebound will be calculated, measured as the TR divided by the time from temperature nadir to temperature peak. This will be termed: temperature rebound rate (TRR).

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Cahill, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nanda S, Levin V, Martinez MW, Freudenberger R. Ranolazine--treatment of ventricular tachycardia and symptomatic ventricular premature beats in ischemic cardiomyopathy. Pacing Clin Electrophysiol. 2010 Dec;33(12):e119-20. doi: 10.1111/j.1540-8159.2010.02733.x. PMID 20345626
- [Background] Deshmukh SH, Patel SR, Pinassi E, Mindrescu C, Hermance EV, Infantino MN, Coppola JT, Staniloae CS. Ranolazine improves endothelial function in patients with stable coronary artery disease. Coron Artery Dis. 2009 Aug;20(5):343-7. doi: 10.1097/MCA.0b013e32832a198b. PMID 19444092
- [Background] Sossalla S, Wagner S, Rasenack EC, Ruff H, Weber SL, Schondube FA, Tirilomis T, Tenderich G, Hasenfuss G, Belardinelli L, Maier LS. Ranolazine improves diastolic dysfunction in isolated myocardium from failing human hearts--role of late sodium current and intracellular ion accumulation. J Mol Cell Cardiol. 2008 Jul;45(1):32-43. doi: 10.1016/j.yjmcc.2008.03.006. Epub 2008 Mar 14. PMID 18439620
- [Background] Gul KM, Ahmadi N, Wang Z, Jamieson C, Nasir K, Metcalfe R, Hecht HS, Hartley CJ, Naghavi M. Digital thermal monitoring of vascular function: a novel tool to improve cardiovascular risk assessment. Vasc Med. 2009 May;14(2):143-8. doi: 10.1177/1358863X08098850. PMID 19366821
- [Background] Kumar K, Nearing BD, Bartoli CR, Kwaku KF, Belardinelli L, Verrier RL. Effect of ranolazine on ventricular vulnerability and defibrillation threshold in the intact porcine heart. J Cardiovasc Electrophysiol. 2008 Oct;19(10):1073-9. doi: 10.1111/j.1540-8167.2008.01204.x. Epub 2008 May 9. PMID 18479333
- [Background] Sicouri S, Glass A, Belardinelli L, Antzelevitch C. Antiarrhythmic effects of ranolazine in canine pulmonary vein sleeve preparations. Heart Rhythm. 2008 Jul;5(7):1019-26. doi: 10.1016/j.hrthm.2008.03.018. Epub 2008 Mar 21. PMID 18598958